CLINICAL TRIAL: NCT06149559
Title: An Open-label, Single-arm Study Evaluating the Activity, Safety, and Pharmacokinetics of Rozanolixizumab in Pediatric Study Participants With Moderate to Severe Generalized Myasthenia Gravis
Brief Title: A Study of Rozanolixizumab in Pediatric Study Participants With Moderate to Severe Generalized Myasthenia Gravis
Acronym: roMyG
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0006; 2022-502074-16-00 (Registry Identifier: CTIS); U1111-1285-0787 (Other: Universal Trial Number)
Record Dates: First submitted 2023-09-25; First posted 2023-11-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Generalized Myasthenia Gravis; gMG; rozanolixizumab; pediatric
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- rozanolixizumab (Experimental): Study participants will receive pre-defined doses of rozanolixizumab for 6 weeks.
  Interventions: Drug: rozanolixizumab

INTERVENTIONS:
Drug: rozanolixizumab — rozanolixizumab solution for injection
  Other Names: UCB7665

SUMMARY:
The purpose of the study is to assess the safety and tolerability of subcutaneous (sc) administration of rozanolixizumab in pediatric participants aged ≥2 to <18 years with generalized Myasthenia Gravis (gMG).

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥2 to <18 years of age inclusive, at the time of signing the informed consent/assent according to local regulation
* Study participant must have a documented diagnosis of generalized Myasthenia Gravis (gMG) at Screening that includes a record confirming the presence of MG specific autoantibodies to acetylcholine receptor (AChR) or muscle-specific kinase (MuSK) prior to Screening
* Study participant has Myasthenia Gravis Foundation of America (MGFA) Clinical Classification II to IVa at Screening
* Study participant has received existing conventional treatment(s) for gMG (eg, pyridostigmine, corticosteroids, and/or immune suppressants) prior to Screening
* Study participant has had an unsatisfactory clinical response or worsening of gMG symptoms and is in need of additional therapy (for example, plasma exchange (PEX) or treatment with intravenous immunoglobulin (IVIg))

Exclusion Criteria:

* Study participant with severe weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis at Screening or Baseline
* Study participant has a known hypersensitivity to any components of the Investigational Medicinal Product (IMP) or other anti-neonatal-Fc receptor (FcRn) medications
* Study participant with any active or untreated thymoma
* Study participant has a history of thymectomy within 6 months prior to Screening
* Study participant has a clinically relevant active infection (eg, sepsis, pneumonia, or abscess) in the opinion of the Investigator, or had a serious infection (resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to the first dose of IMP
* Study participant has received a live vaccination within 4 weeks prior to Baseline or intends to have a live vaccination during the course of the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-06-08 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Occurrence of serious Treatment-Emergent Adverse Events (TEAEs) up to the End of Study (EOS) Visit | From Baseline up to the EOS Visit (up to 18 weeks)
  Serious TEAEs are any untoward medical incidence in a subject during administered study treatment, whether or not these events are related to study treatment and additionally are emergent untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalisation or prolongation of existing hospitalisation
  * Results in persistent disability/incapacity
  * Is a congenital anomaly or birth defect
  * Important medical events
Occurrence of TEAEs leading to permanent withdrawal of Investigational Medicinal Product (IMP) up to the EOS Visit | From Baseline up to the EOS Visit (up to 18 weeks)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Occurrence of Adverse Event(s) of Special Monitoring (AESM) up to the EOS Visit (up to 18 weeks) | From Baseline up to the EOS Visit (up to 18 weeks)
  AESMs are: Severe and/or serious headache, suspected aseptic meningitis, severe Gastrointestinal (GI) disorders, and opportunistic infection.

SECONDARY OUTCOMES:
Percent change in total Immunoglobulin G (IgG) from Baseline at the end of Week 6 | From Baseline to the end of Week 6
  Plasma concentration analyses of total IgG will be done for all study participants on an ongoing basis throughout the study.
Absolute change in total IgG from Baseline at the end of Week 6 | From Baseline to the end of Week 6
  Plasma concentration analyses of total IgG will be done for all study participants on an ongoing basis throughout the study.
Percent change from Baseline in myasthenia gravis (MG) autoantibody levels at the end of Week 6 | From Baseline to the end of Week 6
  Plasma concentration analyses of MG specific anti-acetylcholine receptor (AChR) or anti-muscle-specific kinase (MuSK) autoantibodies will be done for all study participants on an ongoing basis throughout the study.
Absolute change from Baseline in MG-specific autoantibody levels at the end of Week 6 | From Baseline to the end of Week 6
  Plasma concentration analyses of anti-AChR or anti-MuSK autoantibodies will be done for all study participants on an ongoing basis throughout the study.
Change from Baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) total score at the end of Week 6 | From Baseline to the end of Week 6
  The MG-ADL score is an 8-item patient-reported outcome (PRO) instrument. The MG-ADL targets symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The item responses are scored from 0 to 3, and the total score of MG-ADL is the sum of the 8 items and ranges from 0 to 24, with a higher score indicating more disability.
Change from Baseline in Quantitative Myasthenia Gravis (QMG) total score at the end of Week 6 | From Baseline to the end of Week 6
  QMG score is a standardized and validated quantitative strength scoring system that was developed specifically for MG. The QMG total score is obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity.
Occurrence of other TEAEs (including headache, nausea, and infusion site reactions) during Treatment Period 1 (TP1) and Observation Period 1 (OP1) | During TP1 and OP1 (up to 14 weeks)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Evaluation of local tolerability at each scheduled assessment during TP1 | At each scheduled assessment during TP1 (Baseline, week 2, 3, 4, 5, up to 6 weeks)
  Local tolerability will be evaluated at each scheduled assessment for all study participants during TP1.
Plasma concentration of rozanolixizumab at the 6-week treatment cycle | At the 6-week treatment cycle
  Plasma concentration analyses of rozanolixizumab will be done for all study participants on an ongoing basis throughout the study.
Incidence of antidrug antibodies (ADAs) at the end of Week 6 | At the end of Week 6
  Plasma concentration analyses of ADAs will be done for all study participants on an ongoing basis throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (12):
- Mg0006 50574, Denton, Texas, United States
- Italy (3):
  - Mg0006 40290, Bologna
  - Mg0006 40144, Milan
  - Mg0006 40733, Napoli
- Japan (3):
  - Mg0006 20340, Fuchu-shi
  - Mg0006 20339, Ōbu
  - Mg0006 20343, Sagamihara
- Poland (2):
  - Mg0006 40734, Lodz
  - Mg0006 40155, Warsaw
- Taiwan (2):
  - Mg0006 20081, Taipei
  - Mg0006 20095, Taipei
- Mg0006 40836, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org